CLINICAL TRIAL: NCT05437523
Title: A Revolutionary Approach to Managing Functional Constipation in Children Using Digital Education Videos, and Personalized Constipation Action Plans
Brief Title: Clinical Implementation of a Pictographic Constipation Action Plan for Children With Functional Constipation
Acronym: USCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-EDO-2020-0443, 921062
Record Dates: First submitted 2022-06-14; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Functional Constipation
Keywords: clinical action plan
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Toilet-trained children aged four years and older were enrolled if they were evaluated in our institution's pediatric gastroenterology clinic and were diagnosed with functional constipation based on the ROME IV criteria.
  Children were excluded if they were expected to have alternative ROME IV diagnoses (e.g., irritable bowel syndrome), or if an alternative etiology was suspected to be a cause of their constipation.
  Subjects were then block randomized to either receive a constipation action plan or the standard of care (control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group participants received a constipation action plan (USCAP) (Experimental): Received a personalized, pictographic, constipation action plan which detailed the subjects medications to manage functional constipation. The action plan was downloaded from:
  https://wrnmmc.libguides.com/pediatrics/USAP
  Watched a study group, specific, education video. Followed up in 4 months.
  Interventions: Other: Constipation Action Plan
- Control (Active Comparator): Received medications to treat functional constipation Did not receive a written action plan. Watched a control group, specific, education video. Followed up in 4 months.
  Interventions: Other: Standard of care without constipation action plan

INTERVENTIONS:
Other: Constipation Action Plan — The author team previously developed and assessed this constipation action plan using the universal precautions approach to produce a tool which could optimize knowledge transfer from clinicians to patients, and support stepwise home self-management of functional constipation. The Uniformed Services Constipation Action Plan can be freely downloaded at the following web link: https://wrnmmc.libguides.com/pediatrics/USAP
  Arms: Study group participants received a constipation action plan (USCAP)
Other: Standard of care without constipation action plan — Standard of care without constipation action plan
  Arms: Control

SUMMARY:
Constipation is a common disorder that globally affects 0.7% to 29.6% of children. The majority of these children receive the diagnosis of functional constipation. Functional Constipation can be challenging to diagnose and treat. The ROME IV criteria provides structure in the approach to Functional Constipation by standardizing diagnosis criteria. Functional Constipation should be suspected when a child has at least two symptoms per week for the last month consisting of: two or fewer defecations in the toilet per week, greater than or equal to 1 episode of fecal incontinence per week, history of retentive posturing or excessive volitional stool retention, history of painful or hard bowel movements, presence of a large fecal mass in the rectum, or history of large diameter stools that can obstruct the toilet.

Written action plans and similar self-management tools have been associated with improved clinical and patient-reported outcomes for several pediatric chronic disease processes including anaphylaxis, asthma, and atopic dermatitis. These tools have been shown to improve patient/caregiver confidence in disease self-management at home, to increase adherence to pharmacotherapy regimens, and ultimately to enhance patient-centered outcomes. The impact of a Constipation Action Plan on Functional Constipation clinical and patient-related outcomes has not been investigated. The aim of this project was to implement and to evaluate the effectiveness of the Uniformed Services Constipation Action Plan in the management of children with Functional Constipation in a pediatric gastroenterology clinic.

DETAILED DESCRIPTION:
Bakcground

Worldwide, it is estimated that constipation affects 0.7% to 29.6% of children. Constipation accounts for 3% to 10% of general pediatric outpatient visits and up to 25% of visits to pediatric gastroenterologists. Constipation is often associated with infrequent and/or painful defecation, fecal incontinence, and abdominal pain. Furthermore, it may result in significant distress to the child and family, and has a significant impact on health care cost, school absenteeism, and parental workdays missed. While there are concerning organic causes of constipation, - the diagnosis for the 90% of pediatric constipation complaints is not attributable to an organic etiology and is thus classified as functional.

When a child meets these criteria, the diagnosis of functional constipation can be made when, after appropriate evaluation is performed, the patient's symptoms cannot be fully explained by another medical condition.

Multiple research investigations have demonstrated the negative effects on quality of life of pediatric patients with functional constipation as well as the negative effect of this diagnosis on their parents and other caregivers. This impaired health related quality of life (HRQoL) exhibited by children with constipation is lower not only than those of healthy controls, but also lower than children with other significant gastrointestinal diseases such as inflammatory bowel disease or gastroesophageal reflux disease.

In 2014, the pediatric gastroenterology team from Boston Children's Hospital began to advocate for a new "Shared Care" model which implemented of a collaborative quality improvement plan by coordinating a special education program for surrounding primary care managers (PCM) with a focus on the diagnosis and management of functional constipation in children. After developing a constipation management algorithm, The Boston Children's team would conduct digital education with PCMs to discuss constipation pathophysiology as well as the application of the Boston Children's constipation management algorithm. Post-intervention analysis revealed decreased referrals to the pediatric gastroenterology service, which was attributed to improved provider education.

Beyond empowering providers in the chronic care of children, there are multiple examples of other novel interventions to empower patients and parents to better manage chronic conditions, when away from the Patient Centered Medical Home.

Specifically, clinical symptom action plans including those for constipation, asthma, anaphylaxis, and eczema have all been used in the clinical arena. These plans are tailored specifically to the medical needs of the have demonstrated the ability to decrease hospital admissions, decrease emergency department visits, and improve satisfaction for home care by parents. Of note, investigators at the Albert Einstein Colle of Medicine have shown that the implementation of an asthma action plan program decreases hospital admissions, decreases emergency department visits, and decreases medical resource cost.

While appropriate pharmacotherapy and the use of constipation action plans have demonstrated varying scientific rigor within the literature, current clinical practice guidelines and available evidence fail to address the root of the constipation problem in children- which include lifestyle factors such as diets low in fiber, inadequate hydration, poor posturing and other maladaptive behaviors. Direct patient education is key to help address and overcome these obstacles. Most recently a clinical questionnaire for children has placed an emphasis on the clinical impact of behaviors and posturing with the release of the Rome IV Questionnaire for Pediatric Functional gastrointestinal Disorders.

Prior to this, however, current clinical practice guidelines and action plans for constipation have failed to address what many gastroenterologists would consider the root of the constipation problem- poor posturing. The effect of inappropriate straight posturing on the puborectalis angle and the detrimental effect it can have on defecation. The puborectalis muscles acts like a sling encircling the lower colon. When the back is straight and the knees are below the level of the abdomen, the puborectalis muscle contracts causing the colon to kink, thereby impeding the evacuation of stool. When the angle is changed by lifting the knees higher, an angle of 35 degrees can be attained which has been associated with decreased constipation in adults. As a standard of care, posture modification has been made possible through the use of a Defecation Posture Modification Device (DPMD). As a minimal-cost, non-pharmacologic means of therapy, the DPMD is postured to enact real change on the care of constipation in children by serving as a stool for children to prop their feet on and achieve the desired 35 degree angle. This along with other behavioral modifications included in the standard of care: sticker charts, scheduled toilet time, and rewards systems may capture the psychological aspect of functional constipation management which warrants additional investigation.

In summary, investigators seek to create a program which combines improved patient/ provider education, incorporates constipation action plans, to shift the care paradigm to rely more intentionally on written clinical action plans to address low health literacy and improve outcomes.

Methods Investigators measured clinical and patient-related outcomes during this quality improvement project.

At the time of enrollment, participants (or a parent proxy) responded to a health literacy questionnaire: The Newest Vital Sign. This enrollment survey also offered use of a defecation posture modification device (DPMD) to participants at no cost. The remainder of the enrollment survey gathered baseline measurements using validated instruments developed for clinical, patient-related, and health confidence outcomes which would be trended over time to grade USCAP effectiveness. These instruments are discussed in greater detail below. Four months later, participants responded to a second survey which repeated these clinical, patient-related, and health confidence measures.

The 4-month study period was selected based on our institutional practice pattern and to capture recurrences in constipation that can occur after the discontinuation of pharmacotherapy following shorter treatment durations outlined in the North American Society for Pediatric Gastroenterology Hepatology and Nutrition (NASPGHAN) clinical practice guideline. Survey 2 used common, real-world, clinically relevant questions to assess for pharmacotherapy adherence. Investigators used two questions adapted from the Self-Report Measure for Medication Adherence from Wilson et al. In order to assess adherence both qualitatively and quantitatively, participants were asked, "How often does the patient take his/her constipation medicine in the way he/she is supposed to?" using the 5-point Likert scale (0- Never, 1- Almost Never, 2-Sometimes, 3-Often, 4-Almost Always). Next, participants responded to the question, "How many months did the patient take their constipation medicines for?" using a continuous rating from 0 to 4 months. Finally, participants were asked if they used a DPMD with every bowel movement.

Measurements of Implementation Effectiveness Investigators evaluated the effectiveness of the USCAP through multiple approaches. These include clinical, adherence, patient-related, and health confidence outcomes. Toilet-trained subjects, aged ≥4 years, who met the ROME IV criteria for FC were block randomized to receive either the USCAP or control. All discharge instructions were to continue pharmacotherapy for 4 months. Investigators measured subjects at enrollment and 4 months. Metrics included: clinical outcomes using the ROME IV Pediatric Diagnostic Questionnaire, patient-related outcomes using the PedsQL™ Gastrointestinal Symptoms Module [PedsGIQL] (a 5-point Likert scale: 0- Never, 1- Almost Never, 2- Sometimes, 3-Often, 4-Almost Always). The PedsGIQL was administered to participants on at the start of the project after the clinic visit concluded, and 4 months after initial visit. The goal was to demonstrate an improvement in HRQoL. HRQoL responses were stratified by calculating Total Scale Scores. Higher Total Scale Scores demonstrated less (fewer) gastrointestinal symptoms and thus higher (better) gastrointestinal-specific HRQoL. Total Scale Scores were calculated by taking the sum of the reverse-scored items and then dividing by the number of items responded to. Finally, self-efficacy using the Health Confidence Score [HCS] (4-point Likert scale: 3-strongly agree, 2-agree, 1-neutral, 0-disagree).

DATA ANALYSIS Treatment success rates of the treatment and control groups (i.e., the proportion of each group which no longer met the definition of functional constipation) were compared at project conclusion. Investigators also performed an analysis to determine the proportion of subjects with self/parent-proxy reported Pediatric Bristol Stool Form Scale (PBSFS) 3 or 4 achieved at the close of the project and the changes in rates of fecal incontinence (FI). Investigators compared Total Scale Scores from the PedsGIQL between treatment and control groups to determine whether significant change occurred during the project. Changes in HCS were analyzed to compare whether the USCAP is associated with higher, sustained health-confidence compared to control. Univariate analyses were conducted using the Kolmogorov-Smirnov test to investigate potential outliers and normality of the data. When continuous variables were found to be normally distributed, values were summarized using means and standard deviations (SD). When data were found to be skewed or non-normal data were summarized with medians and interquartile ranges (IQR). When comparing continuous variables between groups either a Student's t-test or Wilcoxon rank sum tests were used. Frequency data were reported as counts and percentages. Chi-square was used for all categorical comparisons. When any condition had N ≤5, a Fisher's Exact Test was applied. A P-value <0.05 was considered statistically significant. SAS 9.4 (SAS Institute, Cary, NC) was used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Toilet-trained children aged four years and older
* Participants were diagnosed with functional constipation based on the ROME IV criteria

Exclusion Criteria:

* Participants diagnosed with an alternative ROME IV diagnosis (e.g., irritable bowel syndrome)
* Participants diagnosed with an alternative etiology (i.e., organic etiology) to be a cause of their constipation.

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes- ROME IV Pediatric Diagnostic Questionnaire to diagnose Functional Constipation- Start of Study | At the start of the study
  The measure of implementation effectiveness was clinical: whether the subject met the ROME IV criteria for functional constipation based on the Rome IV Diagnostic Questionnaire for Pediatric Gastrointestinal Disorders for Children and Adolescents (ROME IV Pediatric Diagnostic Questionnaire).
  Scoring instructions for Functional Constipation:
  Two or more of the following:
  (C 1) Two or fewer stools per week, OR (C3) painful stool] OR (C4) Passage of very large stools, OR (C5) Stool retention "once a week" or more often, OR (C6) History of large fecal mass in rectum, OR (C7) Soiling "once a week" or more often.
Clinical outcomes- ROME IV Pediatric Diagnostic Questionnaire to diagnose Functional Constipation- End of Study | At the end of the study (4-months after study start)
  The measure of implementation effectiveness was clinical: whether the subject met the ROME IV criteria for functional constipation based on the Rome IV Diagnostic Questionnaire for Pediatric Gastrointestinal Disorders for Children and Adolescents (ROME IV Pediatric Diagnostic Questionnaire).
  Scoring instructions for Functional Constipation:
  Two or more of the following:
  (C 1) Two or fewer stools per week, OR (C3) painful stool] OR (C4) Passage of very large stools, OR (C5) Stool retention "once a week" or more often, OR (C6) History of large fecal mass in rectum, OR (C7) Soiling "once a week" or more often.
Patient-related outcomes-PedsQL™ Gastrointestinal Symptoms Version 3.0 (PedsGIQL) | start the 4-month study
  Patient-related outcomes were measured using the PedsQL™ Gastrointestinal Symptoms Version 3.0 (PedsGIQL).
  The PedsGIQL includes 11 domains (76 questions): stomach pain, stomach upset, food and drink limits, trouble swallowing, heartburn and reflux, gas and bloating, constipation, diarrhea, worry, medicines, and communication.
  The questions are all graded on 5-point Likert scales (0- Never, 1- Almost Never, 2-Sometimes, 3-Often, 4-Almost Always). Once items were recorded, all items were reverse-scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0) to calculate Total Scale Scores per instructions from Varni (the creator of the tool).
  Higher Total Scale Scores demonstrated less (fewer) gastrointestinal symptoms and thus higher (better) gastrointestinal-specific healthcare related quality of life.
Patient-related outcomes-PedsQL™ Gastrointestinal Symptoms Version 3.0 (PedsGIQL) | end of the 4-month study
  Patient-related outcomes were measured using the PedsQL™ Gastrointestinal Symptoms Version 3.0 (PedsGIQL).
  The PedsGIQL includes 11 domains (76 questions): stomach pain, stomach upset, food and drink limits, trouble swallowing, heartburn and reflux, gas and bloating, constipation, diarrhea, worry, medicines, and communication.
  The questions are all graded on 5-point Likert scales (0- Never, 1- Almost Never, 2-Sometimes, 3-Often, 4-Almost Always). Once items were recorded, all items were reverse-scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0) to calculate Total Scale Scores per instructions from Varni (the creator of the tool).
  Higher Total Scale Scores demonstrated less (fewer) gastrointestinal symptoms and thus higher (better) gastrointestinal-specific healthcare related quality of life.
Health confidence- Health Confidence Score to measure self-efficacy- Start of Study | measured using validated questionnaire at the start of the 4-month study
  Health confidence for home management of functional constipation was measured using the Health Confidence Score (HCS), a tool with established external validity for chronic disease self-management.
  The HCS is a low HL health confidence inventory assesses health knowledge, capability to self-manage, access to help, and shared decision-making using a 4-point Likert scale with pictographs (3-strongly agree, 2-agree, 1-neutral, 0-disagree).
  Higher scores correspond to higher (i.e., better) health confidence.
Health confidence- Health Confidence Score to measure self-efficacy- End of Study | measured using validated questionnaire at the End of the 4-month study
  Health confidence for home management of functional constipation was measured using the Health Confidence Score (HCS), a tool with established external validity for chronic disease self-management.
  The HCS is a low HL health confidence inventory assesses health knowledge, capability to self-manage, access to help, and shared decision-making using a 4-point Likert scale with pictographs (3-strongly agree, 2-agree, 1-neutral, 0-disagree).
  Higher scores correspond to higher (i.e., better) health confidence.

SECONDARY OUTCOMES:
medication adherence, 1 of 2 outcomes measure for Adherence | at end of 4-month study
  Investigators used two questions adapted from the Self-Report Measure for Medication Adherence from Wilson et al. to assess adherence. For the first adherence measure, participants were asked, "How often does the patient take the constipation medicine in the way is supposed to?" using the 5-point Likert scale (0- Never, 1- Almost Never, 2-Sometimes, 3-Often, 4-Almost Always).
  Higher scores correspond to higher (i.e., better) medication adherence.
medication adherence, 2 of 2 outcomes measure for Adherence | at end of 4-month study
  Investigators used two questions adapted from the Self-Report Measure for Medication Adherence from Wilson et al. to assess adherence. For the second adherence measure, participants were asked, "How many months did the patient take their constipation medicines for?" using a continuous rating from 0 to 4 months.
  Higher scores correspond to longer (i.e., better) medication adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IRB did not approve an IPD

REFERENCES:
- [Background] Reeves PT, Kolasinski NT, Yin HS, Alqurashi W, Echelmeyer S, Chumpitazi BP, Rogers PL, Burklow CS, Nylund CM. Development and Assessment of a Pictographic Pediatric Constipation Action Plan. J Pediatr. 2021 Feb;229:118-126.e1. doi: 10.1016/j.jpeds.2020.10.001. Epub 2020 Oct 15. PMID 33068567
- See also: Related Info — https://wrnmmc.libguides.com/pediatrics/USAP